CLINICAL TRIAL: NCT00919659
Title: Parenteral Nutrition Support for Patients With Pancreatic Cancer. A Phase II Study.
Brief Title: Parenteral Nutrition Support for Patients With Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CONKO-Studiengruppe (Other)
Collaborators: Fresenius AG (Industry)
Responsible Party: Helmut Oettle MD, Universitätsmedizin Berlin - Charité
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: C25.0
Record Dates: First submitted 2009-06-09; First posted 2009-06-12 (Estimated); Last update posted 2009-06-12 (Estimated); Status verified 2009-06

CONDITIONS: Cancer Cachexia; Pancreatic Cancer
Keywords: parenteral nutrition; cancer cachexia; pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Hyperphagia | interventions — Parenteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- parenteral nutrition (Experimental): 25kcal/kg/bw /day via parenteral support
  Interventions: Dietary Supplement: parenteral nutrition

INTERVENTIONS:
Dietary Supplement: parenteral nutrition — 25kcal/kg bw with parenteral nutrition
  Other Names: no specific brand name

SUMMARY:
The purpose of this study is to determine whether the additional nutrition support is improving the nutritional status of patients suffering cancer caxechia or not.

DETAILED DESCRIPTION:
To examine the impact of additional parenteral nutrition (APN) we prospective evaluated 32 pts suffering APC and progressive cachexia. This assay is based on a bioelectrical impedance analysis (BIA) as a proven tool for nutritional investigation in patients with chronic disease. Phase angle, determined by BIA, has been found to be a prognostic indicator in several chronic and malignant conditions, such as HIV, liver cirrhosis, chronic obstructive pulmonary disease lung cancer and pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* histological proved pancreatic cancer
* progressive cancer cachexia
* refractive to enteral supplementation
* informed consent

Exclusion Criteria:

* prefinal status
* septic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2002-01; Primary Completion 2004-01 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
nutritional status presented by phase angle | 12 weeks

SECONDARY OUTCOMES:
quantity of port infections, quantity of oedema, quantity of diarrhea | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: helmut oettle, MD, Principal Investigator — CONKO-Studiengruppe
Locations (1):
- Universitätsmedizin Berlin - Charité, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Pelzer U, Arnold D, Govercin M, Stieler J, Doerken B, Riess H, Oettle H. Parenteral nutrition support for patients with pancreatic cancer. Results of a phase II study. BMC Cancer. 2010 Mar 9;10:86. doi: 10.1186/1471-2407-10-86. PMID 20214798